CLINICAL TRIAL: NCT05793346
Title: Pregnancy-associated Progression of Chronic Kidney Disease: A Study Protocol for the Development and Validation of a Clinical Predictive Tool
Acronym: PREDICT
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: King's College London (Other)
Responsible Party: Sponsor
Other Study IDs: PREDICT_Protocol_V1
Record Dates: First submitted 2023-03-06; First posted 2023-03-31 (Actual); Last update posted 2023-03-31 (Actual); Status verified 2023-03

CONDITIONS: Chronic Kidney Diseases; Pregnancy Related
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Dataset 1: National Registry of Rare Kidney Diseases: This dataset is the: National Registry of Rare Kidney Diseases from the UK Renal Registry, this is a UK-wide, linked dataset. This cohort includes any woman who has previously had a previous diagnosis of kidney disease in the UK with maternity records and who has consented to participate.
- Dataset 2: Kent Integrated Data: Maternal and laboratory data from East and West Kent in the UK.
- Dataset 3: Stockholm Creatinine Measurement: An observational dataset with laboratory data from individuals in Stockholm (Sweden)
- Dataset 4: Ontario Renal Network Pregnancy Cohort: A population-based cohort of women in Ontario who had an obstetric delivery with outpatient laboratory data.
- Dataset 5: Combined cohort of three obstetric studies within the UK: A combined cohort derived from three obstetric studies within the UK.

SUMMARY:
To develop and validate a tool that estimates the degree of pregnancy-associated progression of renal disease in women with CKD and pregnancy outcomes in an international multicentre cohort study.

DETAILED DESCRIPTION:
The aim of this study is to develop and validate a tool that estimates the degree of pregnancy-associated progression of renal disease in women with CKD and pregnancy outcomes in an international multicentre cohort study. Two prediction models will be developed to estimate the likelihood of both outcomes. The models will be developed and internally validated in one cohort in the United Kingdom and then externally validated using four international datasets.

ELIGIBILITY:
Inclusion Criteria:

* Women with an estimated Glomerular Filtration Rate (eGFR) using the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) without ethnicity adjustment, less than 90mls/min/1.73m2 within 24 months pre-conception will be included

Exclusion Criteria:

* Women established on dialysis at time of conception
* Multi-fetal pregnancies
* Known inpatient eGFR measurement
* No preconception eGFR within 24 months will be excluded.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Women with pre-existing chronic kidney disease, defined as eGFR < 90mls/min/1.73m2 within 24 months of conception.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2023-03 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Primary outcome a 25% or greater decline in eGFR between six weeks and 12 months postpartum or initiation of dialysis | Six weeks to 12 months postpartum
  A >=25% reduction in eGFR between six weeks and 12 months postpartum or initiation of dialysis.

SECONDARY OUTCOMES:
Secondary outcome: a preterm birth less than 34 weeks or small for gestational age less than 3rd percentile. | To be recorded within 24 hours of date of delivery (Index event is the day of delivery). This outcome is measured on date of delivery.
  A composite outcome of preterm birth defined as less than 34 weeks gestation and/or SGA < 3rd percentile.

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual participant data.

REFERENCES:
- [Background] Wiles K, Webster P, Seed PT, Bennett-Richards K, Bramham K, Brunskill N, Carr S, Hall M, Khan R, Nelson-Piercy C, Webster LM, Chappell LC, Lightstone L. The impact of chronic kidney disease Stages 3-5 on pregnancy outcomes. Nephrol Dial Transplant. 2021 Nov 9;36(11):2008-2017. doi: 10.1093/ndt/gfaa247. PMID 33313680
- [Background] Tong A, Jesudason S, Craig JC, Winkelmayer WC. Perspectives on pregnancy in women with chronic kidney disease: systematic review of qualitative studies. Nephrol Dial Transplant. 2015 Apr;30(4):652-61. doi: 10.1093/ndt/gfu378. Epub 2014 Dec 18. PMID 25523452
- [Background] Piccoli GB, Zakharova E, Attini R, Ibarra Hernandez M, Orozco Guillien A, Alrukhaimi M, Liu ZH, Ashuntantang G, Covella B, Cabiddu G, Li PKT, Garcia-Garcia G, Levin A. Pregnancy in Chronic Kidney Disease: Need for Higher Awareness. A Pragmatic Review Focused on What Could Be Improved in the Different CKD Stages and Phases. J Clin Med. 2018 Nov 5;7(11):415. doi: 10.3390/jcm7110415. PMID 30400594